CLINICAL TRIAL: NCT07400315
Title: A Prospective, Single-arm, Multicenter, Phase II Clinical Study of Iparomlimab and Tuvonralimab (QL1706) in Combination With Modified FLOT Regimen (TFOX) as First-line Treatment for HER2-negative Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: First-line Treatment of Gastric or Gastroesophageal Junction Adenocarcinoma With Dual Immunotherapy Combined With Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-GasC-QIBA-3035
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Gastric or Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric or Gastroesophageal Junction Adenocarcinoma; Iparomlimab and Tuvonralimab Injection; TFOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Drug: Iparomlimab and Tuvonralimab Injection in combination with TFOX

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab Injection in combination with TFOX — Participants enrolled will receive QL1706 (5 mg/kg, Q3W, d1) + docetaxel (50 mg/m², Q3W, d1) + oxaliplatin (100 mg/m², Q3W, d1) + leucovorin (LV) (400 mg/m², Q3W, d1) + 5-fluorouracil (5-FU) (2400 mg/m², Q3W, continuous infusion for 46 hours). The treatment cycle is 21 days, continuing until disease progression, intolerable toxicity, the investigator determines that the participant no longer benefits, the participant withdraws informed consent, QL1706 treatment is completed for 2 years, or other reasons specified in the protocol.Other Name:

SUMMARY:
A prospective, single-arm, multicenter, Phase II clinical study of Apatolimab Tovolimab (QL1706) in combination with modified FLOT regimen (TFOX) as first-line treatment for HER2-negative advanced gastric or gastroesophageal junction adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* 1. The participant voluntarily agrees to participate in this study, signs the informed consent form, and strictly adheres to the requirements of the study protocol.
* 2. Age ≥18 years and ≤75 years at enrollment, regardless of gender.
* 3. Histologically confirmed unresectable locally advanced or metastatic G/GEJ adenocarcinoma, with inclusion criteria specifying HER2- status (HER2+ status defined as IHC3+ or IHC2+ and FISH+).
* 4. No prior systemic treatment for unresectable locally advanced or metastatic G/GEJ adenocarcinoma; previous neoadjuvant and/or adjuvant therapy is acceptable, but all systemic treatments must have been completed at least 12 months prior to the diagnosis of unresectable or metastatic disease.
* 5. At least one measurable tumor lesion according to RECIST 1.1 criteria.
* 6. ECOG PS of 0 or 1.
* 7. Life expectancy ≥3 months.
* 8. Fully recovered from any toxicities related to prior treatments prior to enrollment in the study.
* 9. BMI >18.
* 10. Adequate function of major organs
* 11. Fertile subjects must use appropriate contraception during the study and for 120 days after the end of the study. They must have a negative serum pregnancy test within 7 days prior to enrollment and must not be breastfeeding.

Exclusion Criteria:

* 1. Any unstable systemic disease: including active infection, uncontrolled hypertension, unstable angina, angina that started within the last 3 months, congestive heart failure (New York Heart Association [NYHA] ≥Class II), myocardial infarction within 6 months prior to enrollment, severe arrhythmias requiring medication, or hepatic, renal, or metabolic diseases.
* 2. Symptomatic brain and/or leptomeningeal metastases.
* 3. Known deficiency of dihydropyrimidine dehydrogenase (DPD).
* 4. QT/QTc interval >450 ms for males, >470 ms for females.
* 5. History of other malignancies within 5 years prior to enrollment, with the exception of adequately treated cervical carcinoma in situ, basal cell carcinoma, or squamous cell carcinoma of the skin.
* 6. History of organ transplantation or autologous/allogeneic stem cell transplantation.
* 7. Currently receiving systemic immunotherapy or hormone therapy other than physiologic replacement therapy.
* 8. Other concurrent anti-tumor treatments.
* 9. Known hypersensitivity or allergic reaction to any component of the study treatment.
* 10. Previous exposure to docetaxel or oxaliplatin (except for adjuvant chemotherapy).
* 11. Previous exposure to immune checkpoint inhibitors (e.g., anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies), immune checkpoint agonists (e.g., antibodies targeting ICOS, CD40, CD137, GITR, OX40), or any immunotherapy targeting tumor immune mechanisms.
* 12. Participants with severe bone marrow failure.
* 13. Any disease, metabolic disorder, or physical examination or laboratory findings that suggest contraindications to the study drug or high-risk factors for treatment complications.
* 14. Known or self-reported human immunodeficiency virus (HIV) infection.
* 15. Participants who are HBV or HCV positive.
* 16. Pregnant or breastfeeding.
* 17. Received a live vaccine within 4 weeks prior to the first dose, or plans to receive a live vaccine during the study.
* 18. Participated in any investigational drug treatment or used any investigational device within 4 weeks prior to the first dose.
* 19. Any condition that the investigator believes may pose a risk to the participant receiving the study drug, or may interfere with the evaluation of the study drug, the safety of the participant, or the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Median progression-free survival | 1 year

SECONDARY OUTCOMES:
Objective response rate ,ORR | 1 year
Disease Control Rate | 1 year
Duration Of Response | 1 year
Overall survival ,OS | up to 5 years after treatment discontinuation
12-month survival rate | 12-month
24-month survival rate | 24-month
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | From ICF through 100 days after the last dose of study treatment

IPD SHARING:
Plan to Share IPD: No